CLINICAL TRIAL: NCT02096419
Title: Effect of Continuous Clopidogrel Dosing Targeted After Platelet Function Testing in Acute Coronary Syndrome Patients Undergoing Percutaneous Coronary Intervention With High On-treatment Platelet Reactivity
Brief Title: Continuous Clopidogrel Dose Adjustment in Acute Coronary Syndrome Patients With High On-treatment Platelet Reactivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zagreb (Other)
Collaborators: Clinical Hospital Centre Zagreb (Other); Ministry of Science, Education and Sport, Republic of Croatia (Other Government)
Responsible Party: Principal Investigator, Jure Samardzic, Jure Samardzic M.D., University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108-1081875-1993-1
Record Dates: First submitted 2014-03-19; First posted 2014-03-26 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Acute Coronary Syndrome
Keywords: clopidogrel; platelet reactivity; acute coronary syndrome; tailoring therapy; outcome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (No Intervention): Patients in this group will receive standard clopidogrel dose
- interventional group (Experimental): Patients in the interventional arm will receive clopidogrel dose adjustment to maintain optimal platelet reactivity determined by Multiplate function analyzer (19-46U).
  They will undergo platelet function testing on day 1,2,3,7,30 and month 2,3,6,9 and 12.
  On first two measurements patients will receive up to 2 additional clopidogrel loading doses (600 mg) and put on 150 mg and 75 mg a day if platelet reactivity >18U and <18U, respectively. Maintenance dose will be determined on following measurements - increased by 75 mg if >46U; not changed if 19-46U; decreased by 75 mg if <19U. Minimal dose - 75 mg; maximal dose 300 mg (for patients >70 years 150 mg)
  Interventions: Drug: Clopidogrel dose adjustment

INTERVENTIONS:
Drug: Clopidogrel dose adjustment — Patients in the interventional arm will receive clopidogrel dose adjustment to maintain optimal platelet reactivity determined by Multiplate function analyzer (19-46U).
  They will undergo platelet function testing on day 1,2,3,7,30 and month 2,3,6,9 and 12.
  On first two measurements patients will receive up to 2 additional clopidogrel loading doses (600 mg) and put on 150 mg and 75 mg a day if platelet reactivity >18U and <18U, respectively. Maintenance dose will be determined on following measurements - increased by 75 mg if >46U; not changed if 19-46U; decreased by 75 mg if <19U. Minimal dose - 75 mg; maximal dose 300 mg (for patients >70 years 150 mg)
  Other Names: antiplatelet therapy tailoring
  Arms: interventional group

SUMMARY:
The purpose of this study is to determine whether continuous clopidogrel dose adjustment targeted after platelet function testing improves outcomes during 12 months of follow-up in acute coronary syndrome patients treated with coronary artery stenting and with determined high platelet reactivity on clopidogrel.

DETAILED DESCRIPTION:
Dual antiplatelet therapy (DAPT) with aspirin and P2Y12 receptor antagonists during 12 months presents cornerstone treatment in acute coronary syndrome (ACS) patients undergoing percutaneous coronary intervention (PCI). Clopidogrel is the most widely used P2Y12 inhibitor despite it's limitations that include highly variable P2Y12-receptor inhibition which causes wide interindividual platelet reactivity variability. Since high on-treatment platelet reactivity (HTPR) on clopidogrel is strongly associated with adverse events, antiplatelet therapy tailoring has been vastly investigated to determine whether individualized approach could improve outcomes. In the time of progressive personalized approach to therapy, effective strategies are needed to minimize the risk of ischemic adverse events without increasing the risk for bleeding.

Aim of this study is to investigate whether continuous clopidogrel dose adjustment according to platelet function testing (PFT) using Multiplate® function analyzer (Roche Diagnostics, Mannheim, Germany) could decrease the rate of adverse events in ACS patients treated with PCI and with HTPR during early and late period of DAPT treatment.

Cut off values for HTPR and enhanced platelet response were set according to the consensus statement at >46 U and <19 U, respectively. PFT and therapy tailoring was performed at day 1, 2, 3, 7, 30 and month 2, 3, 6, 9 and 12.

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndrome patients treated with successful PCI
* age 18-80 years
* determined high on-treatment platelet reactivity

Exclusion Criteria:

* continuous postinterventional glycoprotein (GP) IIbIIIa receptor inhibitor infusion
* thrombocytopenia (<150x109/L)
* significant renal insufficiency (creatinine>200 µmol/L)
* anemia (Htc<30%)
* hemorrhagic diathesis
* history of intracranial bleeding or ischemic cerebrovascular insult 6 months before
* major operation 6 weeks before
* concomitant chronic anticoagulation therapy
* age <18 years and >80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
clinical outcome - composite endpoint of total cardiovascular death, non-fatal myocardial infarction, target vessel revascularization and ischemic stroke | 12 months
  Data will be collected during the entire follow up period on interviews and analyzing patient medical data.

SECONDARY OUTCOMES:
number of bleeding events | 12 months
  BARC classification (Bleeding Academic Research Consortium)
  * Type 0: no evidence of bleeding
  * Type 1: bleeding without need for hospitalization or treatment (e.g. bruising, hematoma, nosebleeds, etc.)
  * Type 2: any clinically overt sign of hemorrhage that is actionable but does not meet criteria for type 3, 4 or 5.
  * Type 3: clinical, laboratory, and/or imaging evidence of bleeding, with healthcare provider responses
  * Type 4: Coronary Artery Bypass Graft-related bleeding
  * Type 5: Fatal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Davor Milicic, MD, PhD, Study Chair — University of Zagreb School of Medicine; Jure Samardzic, MD, Principal Investigator — University of Zagreb School of Medicine
Locations (1):
- University Hospital Centre Zagreb, Zagreb, Croatia